CLINICAL TRIAL: NCT03593590
Title: A Multicentre Non-interventional Study to Assess the Real-world Effectiveness of Ocrelizumab in Patients With Relapsing or Primary Progressive Multiple Sclerosis - The MuSicalE STUDY
Brief Title: Non-interventional Study of Ocrelizumab in Participants With Relapsing or Primary Progressive Multiple Sclerosis
Acronym: MuSicalE
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MN39889
Record Dates: First submitted 2018-07-11; First posted 2018-07-20 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ocrelizumab: Participants with relapsing or primary progressive MS receiving ocrelizumab under routine clinical care.
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — Ocrelizumab is administered as an intravenous infusion in accordance with the approved labelling.
  Other Names: Ocrevus

SUMMARY:
This is a multicentre non-interventional study aimed at evaluating the real-world effectiveness and safety of ocrelizumab treatment in participants with relapsing multiple sclerosis (RMS) or primary progressive multiple sclerosis (PPMS), who have been prescribed ocrelizumab as per routine practice. This study will use a comprehensive combination of participant reported outcomes and conventional multiple sclerosis (MS) endpoints that measure clinical domains commonly affected by MS (e.g. fatigue, hand function, gait, cognition), and their impact on employment, activities of daily living, quality of life and healthcare resource utilization. The incidence, type, and pattern of serious adverse events (SAEs), and of adverse events (AEs) leading to treatment discontinuation will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Must have a definite diagnosis of RMS or PPMS and in whom a decision to initiate ocrelizumab has been taken as part of routine clinical practice
* Must be prescribed ocrelizumab in line with the SmPC
* Must have provided signed informed consent
* Must be able and willing to complete the PROs as per clinical practice

Exclusion Criteria:

* Previously treated with ocrelizumab (including phase II, phase III and phase IIIB clinical trials, local trials and investigator initiated study (IIS) as well as a pre-approval access or compassionate use programmes or local registries that are not compatible with the MuSicalE study design)
* Not receiving ocrelizumab in line with the SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with RMS or PPMS undergoing routine clinical care
Sampling Method: Non-Probability Sample
Enrollment: 1710 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
Changes in the overall SymptoMScreen score in participants with RMS | 4 years
  SymptoMScreen is a battery of 7-point Likert scales for 12 distinct domains: mobility, dexterity, body pain, sensation, bladder function, fatigue, vision, dizziness, cognition, depression, and anxiety.
  Composite scores (range min: 0, max: 72) Subscores for each functional domain (range: 0-not affected at all; 6: total limitation/I'm unable to do most daily activities)
Changes in the overall SymptoMScreen score in participants with PPMS | 4 years
  SymptoMScreen is a battery of 7-point Likert scales for 12 distinct domains: mobility, dexterity, body pain, sensation, bladder function, fatigue, vision, dizziness, cognition, depression, and anxiety.
  Composite scores (range min: 0, max: 72) Subscores for each functional domain (range: 0-not affected at all; 6: total limitation/I'm unable to do most daily activities)

SECONDARY OUTCOMES:
Percentage of RMS Participants with Adverse Events | 4 years
Percentage of PPMS participants with Adverse Events | 4 years
Time to treatment discontinuation due to adverse events with ocrelizumab in participants with RMS | 4 years
Time to treatment discontinuation due to adverse events with ocrelizumab in participants with PPMS | 4 years
Change in the score of Multiple Sclerosis Impact Scale (MSIS-29) in RMS participants | 4 years
Change in the score of Multiple Sclerosis Impact Scale (MSIS-29) in PPMS participants | 4 years
Change in the score of ABILHAND - 56 scale in RMS participants | 4 years
Change in the score of ABILHAND - 56 scale in PPMS participants | 4 years
Change in the score of Fatigue Scale Motor and Cognitive functions (FSMC) in RMS participant | 4 years
Change in the score of Fatigue Scale Motor and Cognitive functions (FSMC) in PPMS participants | 4 years
Change in the score of Treatment Satisfaction Questionnaire for Medication (TSQM) in RMS participants | 4 years
Change in the score of Treatment Satisfaction Questionnaire for Medication (TSQM) in PPMS participants | 4 years
Change in the score of MSWS - 12 scale in RMS participants | 4 years
Change in the score of MSWS - 12 scale in PPMS participants | 4 years
Changes in proportion of patients employed/non-employed, number of inpatient days, hospital admissions, medication use and associated costs over the course of the study, captured by the MS-COI in RMS Participants | 4 years
Changes in proportion of patients employed/non-employed, number of inpatient days, hospital admissions, medication use and associated costs over the course of the study, captured by the MS-COI in PPMS Participants | 4 years
Frequency of relapses over time in RMS patients | 4 years
Disease progression in participants with RMS as measured by Expanded Disability Status Scale (EDSS) over time | 4 years
Disease progression in participants with PPMS as measured by Expanded Disability Status Scale (EDSS) over time | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (160):
- Austria (6):
  - Landesklinikum Amstetten, Amstetten
  - Uniklinik fuer Neurologie, Medizinische Universitaet Innsbruck, Innsbruck
  - Kepler Universitätsklinikum GmbH - Neuromed Campus, Linz
  - Kepler Universitätskliniken GmbH - Med Campus III, Linz
  - Multiple Sklerose Zentrum, Melk
  - Klinik Floridsdorf, Vienna
- Belgium (17):
  - Imeldaziekenhuis, Bonheiden
  - AZ KLINA, Brasschaat
  - Hospital Erasme, Brussels
  - UZ Brussel, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - CHU de Charleroi, Charleroi
  - UZ Antwerpen, Edegem
  - CNRF - Centre Neurologique et Réadaptation Fonctionnelle, Fraiture
  - Jessa Zkh (Campus Virga Jesse), Hasselt
  - AZ Groeninge, Kortrijk
  - CHU Tivoli, La Louvière
  - CHC MontLégia, Liège
  - Nationaal MS Centrum, Melsbroek
  - CHU UCL Mont-Godinne, Mont-godinne
  - AZ Oostende, Ostend
  - Revalidatie en MS Centrum, Overpelt
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (5):
  - Clinica Amo - Assistencia Medica Em Oncologia, Salvador, Estado de Bahia
  - Hospital de Base do Distrito Federal, Brasília, Federal District
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - CPQuali Pesquisa Clinica Ltda, São Paulo, São Paulo
  - Hospital Universitario Gaffree e Guinle, Rio de Janeiro
- Bulgaria (11):
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT Sveti Georgi Clinic of neurology, Plovdiv
  - Shat Np Sveti Naum, Sofia
  - First MHAT, Sofia
  - Multiprofile Hosp. for Active Treatment, Sofia
  - "City Clinic UMHAC" EOOD, Sofia
  - Acibadem City Clinic Tokuda Hospital Ead, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT Alexandrovska, EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL EAD, Sofia
  - MBAL St. Marina, Varna
- Clinica Las Condes, Santiago, Chile
- Colombia (4):
  - Fundacion ABOOD Shaio, Bogota, DC
  - Centro Javeriano de Oncología, Bogotá
  - Organizacion Sanitas Internacional, Bogotá
  - Fundacion Clinica Valle del Lili, Cali
- Instituto Nacional del Cáncer Rosa Emilia Sánchez Pérez de Tavares (INCART), Santo Domingo, Dominican Republic
- Egypt (3):
  - Faculty of Medicine-Ain Shams University, Cairo
  - Al Qahira Al Fatmiya Hospital, Cairo
  - Clinical Research Center-Alex university, Cairo
- Italy (24):
  - Ospedale San Salvatore, L’Aquila, Abruzzo
  - Azienda Ospedaliero-Universitaria Consorziale Pol. di Bari, Bari, Apulia
  - Ospedale F. Ferrari, Casarano, Apulia
  - Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - AOU Seconda Università degli Studi, Napoli, Campania
  - Arcispedale Sant'Anna, Cona, Emilia-Romagna
  - A.O.U. di Parma, Parma, Emilia-Romagna
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - Presidio Ospedaliero S.O.P.A. Micone, Sestri Ponente (GE), Liguria
  - Ospedale S.Antonio Abate, Gallarate, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Fond. Istituto Neurologico C.Besta, Milan, Lombardy
  - IRCCS Istituto Neurologico C. Mondino?Dip. Neurologia Neuroriabilitazione S.S. Sclerosi Multipla, Pavia, Lombardy
  - Policlinico San Donato, San Donato Milanese, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
  - Ospedale Regina Montis Regalis, Mondovì (CN), Piedmont
  - Ospedale Binaghi, Cagliari, Sardinia
  - AOU Policlinico V. Emanuele - P.O G. Rodolico, Catania, Sicily
  - AOU Policlinico Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I-G.M. Lancisi-G. Salesi Di Ancona, Torrette - Ancona, The Marches
  - AOU Senese - Presidio Ospedaliero Le Scotte, Siena, Tuscany
- Ibn Sina Hospital, Kuwait City, Kuwait
- Clinical Center of Montenegro, Podgorica, Montenegro
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Maasstadziekenhuis, NL -rotterdam
  - Ziekenhuis VieCuri Medisch Centrum, Venlo
  - Isala, Zwolle
- Hospital Central del Instituto de Previsión Social, Asunción, Paraguay
- Poland (10):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - COPERNICUS Podmiot Leczniczy Sp. z o. o. Szpital im. M. Kopernika, Gdansk
  - Szpital Specjalistyczny im. Swi?tej Rodziny w Rudnej Ma?ej k. Rzeszowa, Głogów Małopolski
  - Gornoslaskie Centrum Medyczne, Katowice
  - UCK im. prof. K. Gibinskiego SUM, Katowice
  - SPZOZ Uniwersytecki Szp. Klin. nr1 im.N.Barlickiego UM, Lodz
  - SPZOZ Wojewodzki Szpital Specjalistyczny nr 3, Rybnik
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Wojskowy Instytut Medyczny - Pa?Stwowy Instytut Badawczy, Warsaw
  - SPSK nr 1, Zabrze
- Portugal (2):
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Centro Hospitalar do Porto, Porto
- Hamad General Hospital, Doha, Qatar
- Romania (5):
  - Fundeni Clinical Institute, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Clinic Judetean de Urgenta Mures, Târgu Mureş
- Russia (4):
  - Jusupovskaya Hospital, Moscow, Moscow Oblast
  - National Center of Social Significant Disease, Saint Petersburg, Sankt-Peterburg
  - Regional clinical hospital named after prof. S.V. Ochapovsky, Krasnodar
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
- King Abdul Aziz Medical City, King Fahd National Guard, Riyadh, Saudi Arabia
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
- Slovakia (6):
  - Univerzitna Nemocnica - Nemocnica svateho Michala, Bratislava
  - Univerzitna nemocnica Bratislava - Nemocnica Ruzinov, Bratislava
  - Nemocnica akademika Ladislava Derera, Bratislava
  - Univerzitna nemocnica Martin, Martin
  - Ustredna vojenska nemocnica SNP Ruzomberok, Ružomberok
  - Fakultna nemocnica Trnava, Trnava
- Spain (24):
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Alava
  - Hospital General Universitario de Elche, Elche, Alicante
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Hospital de Figueres, Figueres, Girona
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Complejo Hospitalario Universitario de Santiago (CHUS) Servicio de Neurologia, Santiago de Compostela, LA Coruna
  - Hospital General Universitario Santa Lucia, Cartagena (Murcia), Murcia
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Nuestra Señora de Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
  - Hospital Universitario Virgen de Arrixaca, Murcia
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Univ. Nuestra Señora de Valme, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
- Turkey (Türkiye) (8):
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul University Istanbul School of Medicine, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Hospital, Kocaeli
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis Univ. Med. Fac., Samsun
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
- Mediclinic Parkview Hospital, Dubai-UAE, United Arab Emirates
- United Kingdom (15):
  - Royal Victoria Hospital, Belfast
  - University Hospital Coventry, Coventry
  - Raigmore Hospital, Inverness
  - Leeds General Infirmary, Leeds
  - Lincoln County Hospital, Lincoln
  - St George?s Hospital, London
  - Luton General Hospital, Luton
  - James Cook Hospital, Middlesbrough
  - John Radcliffe Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Royal Hallamshire Hospital, Sheffield
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - Morriston Hospital, Swansea
  - Southmead Hospital, Westbury-on-Trym, Bristol

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing